CLINICAL TRIAL: NCT03938610
Title: Do Script Concordance Tests Correlate With Family Medicine Standardized Tests and Failing Rotation Grades?
Status: Active, not recruiting | Type: Observational
Sponsor: Pamela Hughes (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Pamela Hughes, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Other Study IDs: FWH20190010H
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Delayed or poor identification and remediation of clinical reasoning difficulties can lead to clinician underperformance and can ultimately compromise patient care. To date, no research has been done to see if SCTs correlate with current grading standards (ITE, ABFM certification exam score, ACGME milestones, or failing clinical rotation grades) in Family Medicine Residents. If investigators can identify that an SCT correlates with current standardized testing of Family medicine residents, it could be possible to identify struggling learners prior to poor scores on the ITE, ACGME milestones, or clinical rotations. If a learner does poorly on an SCT early in the academic year the learner can begin a remediation plan to improve their deficits before receiving a failing grade, poor ITE or ACGME milestone scores.

DETAILED DESCRIPTION:
This study is a longitudinal observation study. A panel of experts (numbering 15-20) consisting of Family Medicine attendings who have been out of residency greater than 3 years will complete the SCT. They will be provided an Informational Consent. Their willingness to be a panel member is their implied consent to be part of the research study.

The basic idea behind SCT is to compare residents' performance with a group of persons who are representatives of the profession (or the specialty) to which they wish to belong. Therefore, panels are made up of physicians with good overall clinical experience in the field rather than experts from narrow parts of the field. Panel composition also depends on the assessment goal.

This study will determine if a Script Concordance Test (SCT) correlates with Family Medicine In Training Exam (ITE) scores, American Board of Family Medicine (ABFM) certification exam scores, Accreditation Council for Graduate Medical Education (ACGME) medical knowledge and patient care milestones, and failing family medicine inpatient clinical rotation grades.

The SCT will be given to PGY1, 2, and 3 residents each year during the Residents three year residency, in June or July.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

--Family Medicine resident at 99MDG

Exclusion Criteria:

-- N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Family medicine residents at 99MDG
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
SCT scores compared to ITE scores | year 1
  SCT scores, ranging from 0 to 100 percent, are longitudinal and will be recorded for all PGY1, 2, and 3 subjects enrolled in the study each year of their residency in June or July.
SCT scores compared to ITE scores | year 2
  SCT scores, ranging from 0 to 100 percent, are longitudinal and will be recorded for all PGY1, 2, and 3 subjects enrolled in the study each year of their residency in June or July.
SCT scores compared to ITE scores | year 3
  SCT scores, ranging from 0 to 100 percent, are longitudinal and will be recorded for all PGY1, 2, and 3 subjects enrolled in the study each year of their residency in June or July.
SCT scores compared to ABFM scores | year 1
  SCT scores, ranging from 0 to 100 percent, are longitudinal and will be recorded for all PGY1, 2, and 3 subjects enrolled in the study each year of their residency in June or July.
SCT scores compared to ABFM scores | year 2
  SCT scores, ranging from 0 to 100 percent, are longitudinal and will be recorded for all PGY1, 2, and 3 subjects enrolled in the study each year of their residency in June or July.
SCT scores compared to ABFM scores | year 3
  SCT scores, ranging from 0 to 100 percent, are longitudinal and will be recorded for all PGY1, 2, and 3 subjects enrolled in the study each year of their residency in June or July.
SCT scores compared to family medicine rotation grades | year 1
  SCT scores, ranging from 0 to 100 percent, are longitudinal and will be recorded for all PGY1, 2, and 3 subjects enrolled in the study each year of their residency in June or July.
SCT scores compared to family medicine rotation grades | year 2
  SCT scores, ranging from 0 to 100 percent, are longitudinal and will be recorded for all PGY1, 2, and 3 subjects enrolled in the study each year of their residency in June or July.
SCT scores compared to family medicine rotation grades | year 3
  SCT scores, ranging from 0 to 100 percent, are longitudinal and will be recorded for all PGY1, 2, and 3 subjects enrolled in the study each year of their residency in June or July.
SCT scores compared to ACGME milestones. | year 1
  SCT scores, ranging from 0 to 100 percent, are longitudinal and will be recorded for all PGY1, 2, and 3 subjects enrolled in the study each year of their residency in June or July.
SCT scores compared to ACGME milestones. | year 2
  SCT scores, ranging from 0 to 100 percent, are longitudinal and will be recorded for all PGY1, 2, and 3 subjects enrolled in the study each year of their residency in June or July.
SCT scores compared to ACGME milestones. | year 3
  SCT scores, ranging from 0 to 100 percent, are longitudinal and will be recorded for all PGY1, 2, and 3 subjects enrolled in the study each year of their residency in June or July.
Binomial SCT classification derived from each interval SCT scores compared to ACGME milestones. | year 1
  A "fail" classification is defined as an SCT score 1 SD below the respective PGY mean. All other SCT scores will be classified as "pass".
Binomial SCT classification derived from each interval SCT scores compared to ACGME milestones. | year 2
  A "fail" classification is defined as an SCT score 1 SD below the respective PGY mean. All other SCT scores will be classified as "pass".
Binomial SCT classification derived from each interval SCT scores compared to ACGME milestones. | year 3
  A "fail" classification is defined as an SCT score 1 SD below the respective PGY mean. All other SCT scores will be classified as "pass".
Binomial SCT classification derived from each interval SCT scores compared to family medicine rotation grades. | year 1
  A "fail" classification is defined as an SCT score 1 SD below the respective PGY mean. All other SCT scores will be classified as "pass".
Binomial SCT classification derived from each interval SCT scores compared to family medicine rotation grades. | year 2
  A "fail" classification is defined as an SCT score 1 SD below the respective PGY mean. All other SCT scores will be classified as "pass".
Binomial SCT classification derived from each interval SCT scores compared to family medicine rotation grades. | year 3
  A "fail" classification is defined as an SCT score 1 SD below the respective PGY mean. All other SCT scores will be classified as "pass".
Binomial SCT classification derived from each interval SCT scores compared to ITE | year 1
  A "fail" classification is defined as an SCT score 1 SD below the respective PGY mean. All other SCT scores will be classified as "pass".
Binomial SCT classification derived from each interval SCT scores compared to ITE | year 2
  A "fail" classification is defined as an SCT score 1 SD below the respective PGY mean. All other SCT scores will be classified as "pass".
Binomial SCT classification derived from each interval SCT scores compared to ITE | year 3
  A "fail" classification is defined as an SCT score 1 SD below the respective PGY mean. All other SCT scores will be classified as "pass".
Binomial SCT classification derived from each interval SCT scores compared to ABFM | year 1
  A "fail" classification is defined as an SCT score 1 SD below the respective PGY mean. All other SCT scores will be classified as "pass".
Binomial SCT classification derived from each interval SCT scores compared to ABFM | year 2
  A "fail" classification is defined as an SCT score 1 SD below the respective PGY mean. All other SCT scores will be classified as "pass".
Binomial SCT classification derived from each interval SCT scores compared to ABFM | year 3
  A "fail" classification is defined as an SCT score 1 SD below the respective PGY mean. All other SCT scores will be classified as "pass".

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Crawford, MD, Study Director — US Air Force
Locations (1):
- Mike O'Callaghan Military Medical Center, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data

REFERENCES:
- [Background] Gagnon R, Charlin B, Coletti M, Sauve E, van der Vleuten C. Assessment in the context of uncertainty: how many members are needed on the panel of reference of a script concordance test? Med Educ. 2005 Mar;39(3):284-91. doi: 10.1111/j.1365-2929.2005.02092.x. PMID 15733164
- [Background] Fournier JP, Demeester A, Charlin B. Script concordance tests: guidelines for construction. BMC Med Inform Decis Mak. 2008 May 6;8:18. doi: 10.1186/1472-6947-8-18. PMID 18460199
- [Background] O'Neill TR, Li Z, Peabody MR, Lybarger M, Royal K, Puffer JC. The Predictive Validity of the ABFM's In-Training Examination. Fam Med. 2015 May;47(5):349-56. PMID 25905876

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT03938610/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT03938610/ICF_001.pdf